CLINICAL TRIAL: NCT05646966
Title: Trunkstability: a Predisposition for Armfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EC2016/0808
Record Dates: First submitted 2017-06-13; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Trunk Stability
Keywords: stroke; reaching; ADL
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy subjects (Active Comparator): healthy subjects
  Interventions: Other: one time testing
- stroke patients (No Intervention): first time stroke patients

INTERVENTIONS:
Other: one time testing
  Arms: healthy subjects

SUMMARY:
Trunk stability is supposed to be an important predisposition for arm function. To the investors knowledge this is never been demonstrated.

DETAILED DESCRIPTION:
Fifty healthy subjects will execute a reaching movement in sitting. They will reach to a cone at a distance of little more than armlength.

Electromyogram (EMG) and kinematics will be the outcome measures. Secondary outcome measures are: sex, dexterity, skillfulness, Fifty first time stroke patients will execute the same movements. Primery outcome is EMG and kinematics; secundary outcome measures are: side of hemiplegia, arm recuperation.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30
* no orthopedic, neurologic disorder that can influence the reaching
* age between 18 and 70 yrs

Exclusion Criteria:

* BMI>30
* orthopedic, neurologic disorder that can influence the reaching
* < 18 yrs of age
* >70 yrs of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Electromyography to analyze muscle activation | 2 hours
  which muscle is active during a reaching movement
kinematics to analyze trunk involvement | 2 hours
  when is the trunk involved in a reaching movement

CONTACTS AND LOCATIONS:
Locations (1):
- Revaki Ugent, Ghent, Oost Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No